CLINICAL TRIAL: NCT05340517
Title: Prospective Study of Video-assisted Rib Planting in Chest Wall Stabilization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weigang Zhao (Other)
Responsible Party: Sponsor-Investigator, Weigang Zhao, Clinical Professor, Shanghai Jiao Tong University Affiliated Sixth People's Hospital
Organization: Shanghai Jiao Tong University Affiliated Sixth People's Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZWG20210222
Record Dates: First submitted 2022-02-14; First posted 2022-04-22 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Rib Fractures; Rib Fracture Multiple
Keywords: internal fixation; video-assisted; chest wall stabilization; prospective study
MeSH Terms: conditions — Rib Fractures | interventions — Thoracic Surgery, Video-Assisted

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- video-assisted rib planting (Experimental)
  Interventions: Procedure: video-assisted rib planting

INTERVENTIONS:
Procedure: video-assisted rib planting — Give the patient intercostal nerve block and laryngeal mask anesthesia, after that, put the patient in lateral position. Make a 4-6cm posterolateral incision along the lower edge of the scapula，sever latissimus dorsi and serratus anterior and reach the rib surface. Lift the scapula with the abdominal retractor (or xiphoid retractor), Free adhesion tissue inside the scapula and put in the thoracoscopic lens. Free the tissue of the upper and lower edges of the ribs carefully, reset ribs and insert rib plate, which is fixed by 90° electric drill and locking screw.
  Other Names: video-assisted thoracoscopic surgery for rib fractures

SUMMARY:
The purpose of this study is to compare the advantages and disadvantages of video-assisted rib planting and traditional internal fixation of rib fractures in chest wall stabilization.

The investigators design a new surgical method of video-assisted thoracoscopic surgery for rib fractures, evaluate the advantages and disadvantages of the new surgical techniques with a prospective study.

ELIGIBILITY:
Inclusion Criteria:

-≥3 unilateral rib displacement fractures

* 18-70 years old
* ASA score I-II
* Preoperative arterial oxygen partial pressure >60mmHg
* Carbon dioxide partial pressure <50mmHg

Exclusion Criteria:

* The distance from the broken end of the posterior rib fracture to the spine is less than 2cm
* Airway stenosis
* Abnormal coagulation system
* History of peptic ulcer or bleeding
* History of allergy to anesthesia related drugs
* History of asthma or chronic obstructive pulmonary emphysema
* Pregnant women

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-02-22 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2022-01-06 (Actual)

PRIMARY OUTCOMES:
The pain score after operation | 6 hours after operation
  The investigators evaluate and record the patients' pain score after operation by visual analog scale (VAS)，which is used to evaluate pain scores 6h,12h,and 24h after the operation.
  0-10 is used to represent different degrees of pain, 0 is painless and 10 is severe pain. The grading criteria of pain were: 0: no pain; 1-3: mild pain; 4-6: moderate pain; 7-10: severe pain.
The pain score after operation | 12 hours after operation
  The investigators evaluate and record the patients' pain score after operation by visual analog scale (VAS).
  0-10 is used to represent different degrees of pain, 0 is painless and 10 is severe pain. The grading criteria of pain were: 0: no pain; 1-3: mild pain; 4-6: moderate pain; 7-10: severe pain.
The pain score after operation | 24 hours after operation
  The investigators evaluate and record the patients' pain score after operation by visual analog scale (VAS).
  0-10 is used to represent different degrees of pain, 0 is painless and 10 is severe pain. The grading criteria of pain were: 0: no pain; 1-3: mild pain; 4-6: moderate pain; 7-10: severe pain.

SECONDARY OUTCOMES:
The postoperative drainage | 7 days at most
  The investigators record the postoperative drainage of patients.The drainage of chest catheter or negative pressure ball was recorded by the nurse every day after surgery.
  Less postoperative drainage means faster recovery and shorter discharge times.

OTHER OUTCOMES:
The operation time | During surgery
  The investigators record patients' operation time duration.
The length of incision | During surgery
  The investigators record the length of operative incision.
The intraoperative bleeding | During surgery
  The investigators record the intraoperative bleeding of patients.
The treatment costs | from the date of hospitalization to the date of leave hospital,assessed up to 100 months
  The investigators record the treatment costs and calculate per capita treatment costs of patients,which is recorded and counted at the time of discharge.
  Total treatment costs include hospitalization, treatment, surgery, medications, and other related expenses.
Days of stay hospital | from the date of hospitalization to the date of leave hospital,assessed up to 100 months
  Days of stay hospital

CONTACTS AND LOCATIONS:
Overall Officials: Weigang Zhao, Principal Investigator — Shanghai Jiao Tong University Affiliated Sixth People's Hospital
Locations (1):
- Shanghai Jiao Tong University Affiliated Sixth People's Hospital, Shanghai, China